CLINICAL TRIAL: NCT02405754
Title: Clinical Utility of an Age, Sex and Gene Expression Score (ASGES or Corus CAD) in the Diagnostic Management of Obstructive Coronary Artery Disease in African American Patients in a Primary Care Setting
Brief Title: Clinical Utility of an Age, Sex, and Gene Expression Score (ASGES or Corus CAD) in African American Patients.
Acronym: AACU
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000024; AACU (Other: CardioDx)
Record Dates: First submitted 2015-03-23; First posted 2015-04-01 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CHD; CVD; CAD
Keywords: Corus CAD; Personalized Medicine; CAD; ASGES; Age/Sex/Gene Expression Score; GES; CVD; CHD; Precision Medicine; Clinical Utility; Gene Expression; Coronary Heart Disease; Cardiovascular Disease; Chest Pain; Coronary Artery Disease; Angina Pectoris; exercise stress testing; CT angiography; invasive cardiac angiography; African-American patient; ICA; CTA
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: Patients receiving Age/Sex/Gene Expression Score (ASGES) or Corus CAD test
  Interventions: Diagnostic Test: Corus CAD (ASGES)

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES

SUMMARY:
This is a retrospective study, designed to be conducted at a single-center in the US. The study will conduct a one-time data abstraction from approximately 500 patient medical charts who received Age/Sex/Gene Expression score (ASGES) also knows as Corus CAD testing, by order of the Principal Investigator. Limited demographic data and patient data pertaining to cardiology referral or advanced diagnostic testing will be collected. All data will be collected anonymously.

DETAILED DESCRIPTION:
Though the diagnostic properties of Age/Sex/Gene Expression Score (ASGES) or Corus CAD have been evaluated in previous observational studies, there are limited data regarding how primary care clinicians are using the results of the test in the care and management of patients with symptoms suggestive of angina in the African-America patient population. This retrospective study is designed to examine the relationship between the Corus CAD (ASGES) score and patterns of care regarding cardiology referral or further cardiac diagnostic testing in an African-American patient population single-center site.

This is a retrospective study, designed to be conducted at a single-center in the US. The study will conduct a one-time data abstraction from approximately 500 patient medical charts who received Corus CAD (ASGES) testing, by order of the Principal Investigator. Limited demographic data and patient data pertaining to cardiology referral or advanced diagnostic testing will be collected. All data will be collected anonymously. IRB approval will be requested with a waiver of informed consent, as no identifying information will be collected.

This retrospective study is designed to understand the patterns of care, including referrals for cardiac care and testing (including referrals to a cardiologist, exercise stress testing, cardiac computerized tomography angiography (CCTA), invasive cardiac angiography (ICA)) within an African-American patient population.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving Corus CAD (ASGES) from 2008-2012.

Exclusion Criteria:

* If any of the following co-moribidities, medical conditions, or current medical statuses are noted in the patient medical chart, s/he will be excluded from the analysis dataset:

  1. History of diabetes;
  2. Revascularization or myocardial infarction;
  3. Systemic infection or inflammatory condition; or
  4. Use of steroids, immunosuppressive agents, or chemotherapeutic agents.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects, who received Age/Sex/Gene Expression Score (ASGES) or Corus CAD testing, will be considered for enrollment by conducting a retrospective review of medical charts. Subjects who satisfy the following inclusion and exclusion criteria will be included for data abstraction.
Sampling Method: Non-Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Referral rate of patients receiving Age/Sex/Gene Expression Score (ASGES) or Corus CAD | Expected follow-up up to 1 year after receiving Corus CAD testing
  Referral rate of patients receiving Age/Sex/Gene Expression Score (ASGES) or Corus CAD , expected follow-up up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ross, MPH, Study Director — CardioDx, Inc.
Locations (1):
- Providence Medical Group - Dayton Primary, Dayton, Ohio, United States